CLINICAL TRIAL: NCT05678309
Title: Establishment of a Patient Library in Patients With Pruritus Sine Materia
Acronym: PRURITHEQUE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC17.0168
Record Dates: First submitted 2022-12-23; First posted 2023-01-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Pruritus; Chronic Pruritus; Itch
MeSH Terms: conditions — Pruritus | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 6 mL of blood will be collected at inclusion to extract the dna
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient library: Patient with pruritus sine materia
  Interventions: Other: Blood samples; Other: skin swab sample; Other: skin biopsy sample; Other: Questionnaires

INTERVENTIONS:
Other: Blood samples — At inclusion :
  * 52.5 ml of blood :
  * 24 ml plasma
  * 20 ml serum
  * 6 ml DNA
  * 2.5 ml RNA
Other: skin swab sample — At inclusion a skin swab sample will be collected
Other: skin biopsy sample — At inclusion a skin biopsy sample will be collected
Other: Questionnaires — At inclusion, at 6 months and every year, the patient will respond to 5 questionnaires : Brest questionnaire, 5-D itch scale, Dermatology Life Quality Index, Itchy Quality of Life and Hospital Anxiety and Depression Scale

SUMMARY:
Very little is currently known about the pathophysiology of pruritus sine materia according to the etiology. The creation of this cohort should make it possible to improve our clinical and biological knowledge according to the etiology, by collecting blood, skin, feces, and clinical data.

DETAILED DESCRIPTION:
At inclusion, 52.5 ml of blood will be collected, then an additional skin biopsy and a skin swab. Five questionnaires will be filled in by the patient.

At 6 months, then every years for 5 years, the same 5 questionnaires will be collected as well as the clinical data. However, no more biological samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pruritus sine materia
* Collection of consent
* Adult

Exclusion Criteria:

- Refusal to participate in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with pruritus sine materia
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical description of the pruritus | 5 years
  Chronology
Clinical description of the pruritus | 5 years
  Intensity
Clinical description of the pruritus | 5 years
  Location
Clinical description of the pruritus | 5 years
  Aggravating and ameliorating factors
Clinical description of the pruritus | 5 years
  Evolution
Clinical description of the pruritus | 5 years
  Scratching
Clinical description of the pruritus | 5 years
  Chronology, intensity, location, aggravating and ameliorating factors, evolution, scratching
5-D itch scale questionnaire | 5 years
  The scores for each of the five domains (duration, degree, direction, disability, ditribution) are calculated separately and then added together to obtain a total 5-D score.
  The 5-D score can range from 5 (no pruritus) to 25 (most severe pruritus). Scores with a single item (duration, degree, direction) are equal to the value indicated by the answer choice (from 1 to 5).
  The impact of pruritus (disability) includes four items that assess the impact of itching on daily activities: sleep, leisure activities, social activities, domestic activities, work/study. The score for impact is reached by taking the highest score on any of the four items.
  For location (distribution), the number of body parts affected is collected (potential sum of 0 to 16) and the sum is classified into 5 scores:
  * sum of 0 to 2 = score of 1
  * sum of 3 to 5 = score of 2
  * sum of 6 to 10 = score of 3
  * sum of 11 to 13 = score of 4
  * sum of 14 to 16 = score of 5
Dermatology Life Quality Index questionnaire (DLQI) | 5 years
  DLQI = Dermatology Life Quality Index is a ten-item questionnaire. The score ranges from 0 to 30. Each question is rated from 0 to 3. The higher the score, the worse the health status.
  Interpretation of DLQI:
  DLQI scores 0-1: no effect on patient's life DLQI scores 2-5: small effect on patient's life DLQI scores 6-10: moderate effect on patient's life DLQI scores 11-20: very large effect on patient's life DLQI scores 21-30: extremely large effect on patient's life
Hospital anxiety and depression questionnaire (HAD) | 5 years
  The HAD scale is an instrument to screen for anxiety and depressive disorders. It consists of 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score = 21).
  To screen for anxiety and depressive symptoms, the following interpretation can be proposed for each of the scores (A and D)
  * 7 or less: no symptomatology
  * 8 to 10: doubtful symptomatology
  * 11 and more: definite symptomatology.
Brest Questionnaire | 5 years
  The Brest questionnaire is a descriptive tool. No score is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de dermatologie, CHRU BREST, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement